CLINICAL TRIAL: NCT02380287
Title: Open-label, Phase I Dose-escalation Clinical Study of the Safety, Tolerability and Pharmacokinetics of Single Subcutaneus Dose of BCD-085, Monoclonal Antibody Against IL-17, in Healthy Subjects
Brief Title: First-in-human Study to Evaluate Safety, Tolerability and Pharmacokinetics of Various Doses of BCD-085 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BCD-085-1
Record Dates: First submitted 2015-03-02; First posted 2015-03-05 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: interleukin-17; maximum tolerated dose; novel monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort no.1 (Experimental): This cohort includes just one subject who will receive the maximum safe starting dose of BCD-085 (0.05 mg/kg) subcutaneously. If the dose limitating toxicity occurs within the first seven days after injection the study will be stopped. If there is no DLT within mentioned above period then Cohort no.2 is included.
  Interventions: Drug: humanized monoclonal antibody against human IL-17
- Cohort no.2 (Experimental): This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-085 at a dose of 0.05 mg/kg.
  If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no. 3 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 3.
  Interventions: Drug: humanized monoclonal antibody against human IL-17
- Cohort no.3 (Experimental): This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-085 at a dose of 0.25 mg/kg.
  If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no. 4 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 4.
  Interventions: Drug: humanized monoclonal antibody against human IL-17
- Cohort no.4 (Experimental): This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-085 at a dose of 0.825 mg/kg.
  If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no. 5 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 5.
  Interventions: Drug: humanized monoclonal antibody against human IL-17
- Cohort no.5 (Experimental): This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-085 at a dose of 1.25 mg/kg.
  If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no. 6 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 6.
  Interventions: Drug: humanized monoclonal antibody against human IL-17
- Cohort no.6 (Experimental): This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-085 at a dose of 1.75 mg/kg.
  If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no. 7 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 7.
  Interventions: Drug: humanized monoclonal antibody against human IL-17
- Cohort no.7 (Experimental): This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-085 at a dose of 2.25 mg/kg.
  If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no. 8 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 8.
  Interventions: Drug: humanized monoclonal antibody against human IL-17
- Cohort no.8 (Experimental): This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-085 at a dose of 3.0 mg/kg.
  If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level.
  Interventions: Drug: humanized monoclonal antibody against human IL-17

INTERVENTIONS:
Drug: humanized monoclonal antibody against human IL-17
  Other Names: BCD-085

SUMMARY:
This is an open label, phase 1, "3+3" dose escalating study of tolerability, safety, pharmacokinetics and immunogenicity of a single subcutaneous injection of the novel monoclonal antibody against human IL-17 - BCD-085. The study will enroll 37 healthy male volunteers.

DETAILED DESCRIPTION:
IL-17 is a new potential therapeutic target which plays important role in pathogenesis of several autoimmune disorders including psoriasis, rheumatoid arthritis, possibly - SLE and MS. BCD-085 is a novel humanized monoclonal antibody against human IL17 developed by JCS BIOCAD (Russia) which is now on the first step of clinical evaluation. BCD-085-1 study is the first-in-human clinical trial which is intended to evaluate tolerability, safety, pharmacokinetics and immunogenicity of BCD-085 when used as a single step-by-step escalating subcutaneous dose in healthy male volunteers. During this study it is expected to determine diapason of safety doses of BCD-085 (incl. MTD) which thereafter can be evaluated in phase 2 studies.

ELIGIBILITY:
Inclusion Criteria:

* singed informed consent
* male gender
* 18-45 years of age inclusively
* BMI between18.5-30.0 kg/sq.m.
* absence of any sings of hepatic, renal, gastrointestinal, cardiovascular, endocrine, respiratory, immunologic, hematologic, dermatologic, or neurologic abnormality at screening or/and in anamnesis
* parameters of complete blood count, blood biochemistry, and urinalysis do not exceed reference values, which are used at Study site laboratory. Evaluation of required laboratory parameters must be performed within 14 days before randomization
* normal hemodynamic parameters : systolic BP 100 - 139 mm Hg, diastolic BP - 60 - 90 mm Hg, heart rate - 60 - 90 b/min
* absence of chronic infections (HIV, syphilis, hepatitis В or С, tuberculosis ) and chronic inflammation
* absence of infections within 4 weeks before randomization
* absence of mental disorders or other conditions (incl. depression), which may affect the ability of participant to follow Protocol
* health well-being (by volunteer's opining opinion) for at least 30 days before randomization.
* absence of alcohol or drug addiction signs (incl. history of such addiction). Consent not to use alcohol within 24 hours before and after injection of BCD-085;
* volunteer's ability to follow Protocol procedures
* consent of volunteers and their sexual partners with childbearing potential to use adequate contraception during screening period and the main study part (14 days before randomization and 61 day after SC injection). This requirement is not applicable in surgically sterilized volunteers. Adequate contraception includes the use of one barrier method in combination with spermicides, intrauterine device / oral contraceptives in sexual partner

Exclusion Criteria:

* history of use of monoclonal antibodies against IL-17
* known severe allergy (anaphylaxis or multidrug intolerance)
* known intolerance to medicines containing monoclonal antibodies (murine, humanized, human) or to any excipients of BCD-085
* major surgery within 30 days prior screening
* severe infections (required hospitalization, parenteral use of antimicrobial agents) within 6 months prior the date of BCD-085 injection
* systemic use of antimicrobials within 2 months prior the date of BCD-085 injection
* more than 4 episodes of respiratory tract infections within 6 months prior the screening examination
* presence of any disorders which may affect pharmacokinetics of BCD-085
* history of fever which was equal or exceeded 40 degrees in Celsius
* history of hepatic transaminases increase 2.5 x ULN
* history of seizures
* actual or prior depression, suicidal tendencies
* use of any medicines, vitamins, biologically active additives within 14 days prior the date of BCD-085 injection
* use of any medicines which affects hemodynamics or hepatic function within 30 days prior the date of BCD-085 injection
* use of any medicines which may influence on immune system within 30 days prior the date of BCD-085 injection
* vaccination within 4 weeks prior the date of BCD-085 injection
* smoking exceeds 10 cigarettes per day
* use of alcohol, which exceeds 10 units per week (1 alcohol unit is equal ½ l of beer (1 pint), or 200 ml of vine, or 50 ml alcohol
* donation of more than 450 ml of blood or plasma within 2 months prior randomization.
* simultaneous participation in any other clinical trial, as well as former participation in other clinical trials within 3 months before this study initiation.
* previous participation in this study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — JCS BIOCAD

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort no.1: This cohort includes just one subject who will receive the maximum safe starting dose of BCD-085 (0.05 mg/kg) subcutaneously. If the dose limitating toxicity occurs within the first seven days after injection the study will be stopped. If there is no DLT within mentioned above period then Cohort no.2 is included.
  humanized monoclonal antibody against human IL-17
- Cohort no.2: This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-085 at a dose of 0.05 mg/kg.
  If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no. 3 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 3.
  humanized monoclonal antibody against human IL-17
- Cohort no.3: This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-085 at a dose of 0.25 mg/kg.
  If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no. 4 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 4.
  humanized monoclonal antibody against human IL-17
- Cohort no.4: This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-085 at a dose of 0.825 mg/kg.
  If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no. 5 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 5.
  humanized monoclonal antibody against human IL-17
- Cohort no.5: This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-085 at a dose of 1.25 mg/kg.
  If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no. 6 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 6.
  humanized monoclonal antibody against human IL-17
- Cohort no.6: This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-085 at a dose of 1.75 mg/kg.
  If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no. 7 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 7.
  humanized monoclonal antibody against human IL-17
- Cohort no.7: This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-085 at a dose of 2.25 mg/kg.
  If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 subjects are observed to have DLT, the dose level is escalated one step for the next cohort no. 8 of 3 subjects, and the process continues as above. If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next Cohort no. 8.
  humanized monoclonal antibody against human IL-17
- Cohort no.8: This cohort includes 3 subjects who will receive the single subcutaneous injection of BCD-085 at a dose of 3.0 mg/kg.
  If at least 2 subjects are observed to have DLT, this dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If exactly 1 of the 3 subjects treated show DLT, 3 additional subjects are treated at the current dose level.
  humanized monoclonal antibody against human IL-17
Period: Overall Study
Arm/Group | Cohort no.1 | Cohort no.2 | Cohort no.3 | Cohort no.4 | Cohort no.5 | Cohort no.6 | Cohort no.7 | Cohort no.8
Started | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 1 | 3 | 2 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort no.1: This cohort includes just one subject who received the maximum safe starting dose of BCD-085 (0.05 mg/kg) subcutaneously.
- Cohort no.2: This cohort includes 3 subjects who received the single subcutaneous injection of BCD-085 at a dose of 0.05 mg/kg.
- Cohort no.3: This cohort includes 3 subjects who received the single subcutaneous injection of BCD-085 at a dose of 0.25 mg/kg.
- Cohort no.4: This cohort includes 3 subjects who received the single subcutaneous injection of BCD-085 at a dose of 0.825 mg/kg.
- Cohort no.5: This cohort includes 3 subjects who received the single subcutaneous injection of BCD-085 at a dose of 1.25 mg/kg.
- Cohort no.6: This cohort includes 3 subjects who received the single subcutaneous injection of BCD-085 at a dose of 1.75 mg/kg.
- Cohort no.7: This cohort includes 3 subjects who received the single subcutaneous injection of BCD-085 at a dose of 2.25 mg/kg.
- Cohort no.8: This cohort includes 3 subjects who received the single subcutaneous injection of BCD-085 at a dose of 3.0 mg/kg.
- Total: Total of all reporting groups
Arm/Group | Cohort no.1 | Cohort no.2 | Cohort no.3 | Cohort no.4 | Cohort no.5 | Cohort no.6 | Cohort no.7 | Cohort no.8 | Total
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 22
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 22

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration of BCD-085-time Curve From Zero (0) Hours to 1344 Hours After the Single Subcutaneous Injection of BCD-085
Description: The blood sampling for the pharmacokinetic evaluations was performed at the following time points: 0 h (5 min before the injection) and at 0.5 hours, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 48 hours, 72 hours,168 hours, 336 hours, 504 hours, 672 hours, 840 hours, 1008 hours, 1176 hours, and 1344 hours following the drug administration.
Time Frame: 56 days
Population: The analysis population includes all subjects for whom not more than 2 blood samples for BCD-085 assay were missing or unevaluable, and for whom no violations of blood sampling schedule were reported. Results of PK parameters consider in Cohort 1 and 2 together since the same dose were injected.
Measure: Median (Inter-Quartile Range); unit: (ng/ml)*hour
Groups:
- Cohort 1 + Cohort 2: This cohort includes subjects who received the single subcutaneous injection of BCD-085 at a dose of 0.05 mg/kg.
- Cohort 3: This cohort includes subjects who received the single subcutaneous injection of BCD-085 at a dose of 0.25 mg/kg.
- Cohort 4: This cohort includes subjects who received the single subcutaneous injection of BCD-085 at a dose of 0.825 mg/kg.
- Cohort 5: This cohort includes subjects who received the single subcutaneous injection of BCD-085 at a dose of 1.25 mg/kg.
- Cohort 6: This cohort includes subjects who received the single subcutaneous injection of BCD-085 at a dose of 1.75 mg/kg.
- Cohort 7: This cohort includes subjects who received the single subcutaneous injection of BCD-085 at a dose of 2.25 mg/kg.
- Cohort 8: This cohort includes subjects who received the single subcutaneous injection of BCD-085 at a dose of 3.0 mg/kg.
Arm/Group | Cohort 1 + Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 4 | 2 | 3 | 3 | 3 | 3 | 3
(ng/ml)*hour | 594222.00 [583105.25 to 597706.25] | 2262670.25 [1600708.75 to 2924631.75] | 5669903.75 [5566847.00 to 7958067.25] | 9939951.75 [8169096.25 to 10963413.25] | 9220825.00 [6191133.50 to 11536130.00] | 14915081.50 [13047990.50 to 14963820.50] | 10152522550.50 [9119054864.00 to 11931556230.00]

2. Secondary Outcome: Maximum Concentration of BCD-085 After Single Subcutaneous Injection
Description: To assess the maximum observed concentration (Cmax) following single SC administer regardless of the cohort
Time Frame: 56 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 + Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 4 | 2 | 3 | 3 | 3 | 3 | 3
ng/mL | 583.5 (53.3) | 2566.00 (504.87) | 8970.67 (1831.26) | 12946.67 (1744.52) | 12415.33 (4280.65) | 20115.00 (1413.55) | 28691.33 (1478.00)

3. Other Pre Specified Outcome: Time of Maximum Concentration of BCD-085 After Single Subcutaneous Injection
Description: To assess the Tmax following single SC administer regardless of the cohort
Time Frame: 56 days
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 + Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 4 | 2 | 3 | 3 | 3 | 3 | 3
hours | 252.000 [168.000 to 336.000] | 168.000 [168.000 to 168.000] | 168.000 [168.000 to 168.000] | 72.000 [72.000 to 72.000] | 48.000 [48.000 to 72.000] | 168.000 [48.000 to 168.000] | 168.000 [168.000 to 336.00]

4. Other Pre Specified Outcome: Half-life of BCD-085 After Single Subcutaneous Injection
Time Frame: 56 days
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 + Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 4 | 2 | 3 | 3 | 3 | 3 | 3
hours | 425.15 [400.20 to 434.86] | 378.78 [349.56 to 408.01] | 370.13 [342.18 to 381.97] | 362.78 [354.71 to 387.87] | 428.42 [410.12 to 448.61] | 370.70 [363.15 to 387.85] | 375.76 [335.11 to 383.68]

5. Other Pre Specified Outcome: Constant of Elimination of BCD-085 After Single Subcutaneous Injection
Time Frame: 56 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours^-1
Arm/Group | Cohort 1 + Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 4 | 2 | 3 | 3 | 3 | 3 | 3
hours^-1 | 0.002 (0.000) | 0.002 (0.000) | 0.002 (0.000) | 0.002 (0.000) | 0.002 (0.000) | 0.002 (0.000) | 0.002 (0.000)

6. Other Pre Specified Outcome: Clearance of BCD-085 After Single Subcutaneous Injection
Time Frame: 56 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Cohort 1 + Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 4 | 2 | 3 | 3 | 3 | 3 | 3
mL/h | 6.18 (2.16) | 10.25 (1.81) | 8.80 (1.04) | 8.75 (2.63) | 16.05 (2.36) | 12.29 (1.43) | 11.45 (1.81)

7. Other Pre Specified Outcome: Mean Pain Score by VAS Assessment During Injection of BCD-085
Description: The study subject assesses how painful was the injection. Assessment is performed by filling out a special 10-score visual analogue scale (VAS) immediately after the injection is done. The 0 score refers to no pain, the score 10 refers to the highest, almost unbearable pain. The pain was assessed after a single injection.
Time Frame: day 1
Population: The safety analysis will include all subjects received BCD-085.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cohort 1: This cohort includes just one subject who received the maximum safe starting dose of BCD-085 (0.05 mg/kg) subcutaneously.
- Cohort 2: This cohort includes subjects who received the same single dose of BCD-085 as in a Cohort 1 (0.05 mg/kg) subcutaneously since no grade 3/4 toxicity events were observed in Cohort 1 during follow-up period (7 days).
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 3
score on a scale | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

8. Other Pre Specified Outcome: Total Frequency of AE/SAE
Time Frame: 56 days
Population: The analysis population includes subjects who received any dose of BCD-085 subcutaneously.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Participants
  Total frequency of AEs | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0
  Total frequency of SAEs | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

9. Other Pre Specified Outcome: Frequency of Local Reactions
Time Frame: 56 days
Population: Safety population included all subjects who received at least one injection of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Other Pre Specified Outcome: Frequency of Grade 3-4 AEs
Time Frame: 56 days
Population: The safety population included all subjects who received at least one injection of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

11. Other Pre Specified Outcome: Frequency of Early Discontinuation Due to AE
Time Frame: 56 days
Population: The safety population included all subjects who received at least one injection of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

12. Other Pre Specified Outcome: Frequency of Binding Antibodies to BCD-85 Formation
Time Frame: day 56
Population: Immunogenicity was evaluated in all volunteers who received the drug administration, and who had both samples, available for analysis. Volunteer from Cohort 3 had early withdrawal, so he did not have a second sample for the study. Thus, the total number of volunteers for immunogenicity assessment was 21.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Cohort no.1 | Cohort no.2 | Cohort no.3 | Cohort no.4 | Cohort no.5 | Cohort no.6 | Cohort no.7 | Cohort no.8
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3 | 1/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/1 | 0/3 | 1/3 | 0/3 | 2/3 | 1/3 | 0/3 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort no.1 (N=1) | Cohort no.2 (N=3) | Cohort no.3 (N=3) | Cohort no.4 (N=3) | Cohort no.5 (N=3) | Cohort no.6 (N=3) | Cohort no.7 (N=3) | Cohort no.8 (N=3)
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort no.1 (N=1) | Cohort no.2 (N=3) | Cohort no.3 (N=3) | Cohort no.4 (N=3) | Cohort no.5 (N=3) | Cohort no.6 (N=3) | Cohort no.7 (N=3) | Cohort no.8 (N=3)
Elevated ALT (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Elevated AST (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No